CLINICAL TRIAL: NCT07062640
Title: The Risk of Sleep Disordered and Dietary Advanced Glycation End Products in Preschool Children
Brief Title: Sleep Quality and dAGE Intake in Preschool Children
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Büşra Demirer, PhD, Karabuk University
Other Study IDs: BD14
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Child Nutrition Disorders
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- sleep disordered: sleep disordered with preschool children
- normal: normal sleep with preschool children

SUMMARY:
The aim was to evaluate the relationship between dietary AGE intake and sleep quality and some nutrient intake of healthy children aged 3-5 years registered in various nurseries in Ankara. The main question that the study aimed to answer is:

Does dietary AGE intake affect sleep quality in preschool children? 304 children (140 girls, 164 boys) were included in the study. According to the SDSC scale, 67.5% of the participants were at risk of sleep disorders. The dAGE intake of children at risk of sleep disorders was significantly higher compared to children with normal sleep status.

ELIGIBILITY:
Inclusion Criteria:

Individuals must be between 3-5 years old

Individuals must participate in the study voluntarily

Individuals must not have cognitive dysfunction

They must be able to answer the survey questions

Exclusion Criteria:

Individuals are not 3-5 years old

Individuals do not want to participate in the study voluntarily

Individuals have cognitive dysfunction

Inability to answer survey questions

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children aged 3-5 registered in various nurseries in Ankara
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-06-13 (Actual)

PRIMARY OUTCOMES:
sleep quality | Baseline
  To categorize sleep disturbances in children, the psychometric properties were evaluated using the 27-item Likert-type rating scale, the SDSC. The total score is 26 - 130. As the score increases, sleep quality deteriorates.
dAGE intake | Baseline
  Dietary AGE measurements were calculated based on the database of Uribarri et al. A 24-hour retrospective food consumption record was obtained from the children.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Demirer, PhD, Principal Investigator — Karabuk University; Gökçen Doğan, PhD, Study Director — Lokman Hekim University; Nurcan Yabancı Ayhan, Prof.Dr., Study Chair — Ankara University
Locations (1):
- Ankara, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No